CLINICAL TRIAL: NCT00919958
Title: Phase I Study of Intramuscular (IM) Injection of Allogeneic PLX-PAD Cells for the Treatment of Critical Limb Ischemia. PLX-PAD Are Mesenchymal-like Stromal Cells Derived From a Full Term Placenta. These Placental Adherent Stromal Cells (ASCs) Are Expanded in the Company's Proprietary PluriXTM 3D Bioreactor System. PLX Cells Are Immune Privileged and Possess Immunomodulatory Properties.
Brief Title: Safety of Intramuscular Injection of Allogeneic PLX-PAD Cells for the Treatment of Critical Limb Ischemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PLX-PAD 1202-1
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease; Critical Limb Ischemia
Keywords: Peripheral Artery Disease; Peripheral Vascular Disease; Critical limb ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PLX-PAD low dose (Experimental)
  Interventions: Biological: PLX-PAD IM injection
- PLX-PAD intermediate dose (Experimental)
  Interventions: Biological: PLX-PAD IM injection
- PLX-PAD high dose (Experimental)
  Interventions: Biological: PLX-PAD IM injection

INTERVENTIONS:
Biological: PLX-PAD IM injection — Single treatment; multiple injections

SUMMARY:
The The purpose of this study is to determine the safety of PLX-PAD single dose, Intra-muscular injection for the treatment of CLI patients.

DETAILED DESCRIPTION:
PLX-PAD are mesenchymal-like stromal cells derived from a full term placenta, termed PLX-PAD, and intended for the treatment of Critical Limb Ischemia

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of critical limb ischemia defined as persistent, recurring ischemic rest pain for at least two (2) weeks, and/or ulceration or gangrene of the foot or toe, with ABI < 0.4 or/and TBI < 0.4 or transcutaneous partial pressure of oxygen ≤ 30 mmHg pO2 at the foot.
2. Rutherford category 4-5
3. No acceptable options for re-vascularisation as confirmed by angiographic imaging results or by color flow duplex ultrasound obtained within 6 months prior screening visit and signed approval of vascular surgeon.
4. In the opinion of the investigator, major amputation is not anticipated over a period of three (3) months.

Exclusion Criteria:

1. Uncontrolled hypertension (defined as diastolic blood pressure > 110 mmHg or systolic blood pressure > 180 mmHg during screening).
2. Poorly controlled diabetes mellitus (HbA1c > 9%)
3. Wounds with severity greater than Grade 2 on the Wagner Scale
4. Life-threatening ventricular arrhythmia - except if an ICD is implanted - or unstable angina pectoris - characterized by increasingly frequent episodes with modest exertion or at rest, worsening severity, and prolonged
5. ST segment elevation myocardial infarction and/or TIA/CVA within six (6) months prior to enrollment. Patients with severe congestive heart failure (i.e. NYHA Stage IV)
6. In the opinion of the investigator, the patient is unsuitable for cellular therapy.

Ages: 40 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Adverse events, Safety laboratory values and ECG findings | 3 months
Immunological reaction | 1 month

SECONDARY OUTCOMES:
Tumorigenesis | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Carsten Tschöpe, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Franziskus-Krankenhaus, Berlin, Germany